CLINICAL TRIAL: NCT01382485
Title: Reamer Irrigator Aspirator Versus Autogenous Iliac Crest Bone Graft for the Treatment of Non-Unions: A Multi-Centre Randomized Controlled Trial
Brief Title: Reamer Irrigator Aspirator (RIA) vs Autogenous Iliac Crest Bone Graft (AICBG) for the Treatment of Non-unions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIA2011
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Nonunion of Bone Graft; Fractures Non Union
Keywords: non union; bone defect; tibia non union; femur non union; bone graft
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AICBG harvesting group (Active Comparator): Iliac crest bone graft will be harvested from the anterior iliac crest through an incision beginning 2cm posterior to the anterior superior iliac spine and carried posteriorly. A window will be made in the iliac crest and a curette will subsequently be used to harvest the cancellous bone. The incision will be closed in 3 layers. The infiltration of local anaesthetic will be at the discretion of the surgeon.
  Interventions: Other: AICBG harvesting group
- RIA harvesting group (Experimental): Subjects allocated to the RIA group will have the graft harvested in a standardized fashion using the technique described by Quintero et al. Briefly, the RIA device is a single-pass reamer that is connected to an aspirator and irrigator, allowing simultaneous reaming, irrigation, and aspiration of the contents of the femoral canal. RIA head size and tube length will be chosen based on preoperative templating of anteroposterior and lateral radiographs of the donor femur (a head size of 2mm larger than the inner cortical diameter at the isthmus of the femur will be selected). Fluoroscopic imaging will be used to confirm guidewire positioning and avoid eccentric reaming. Bone graft will be harvested from the central femoral canal and from each femoral condyle in 3 separate passes.
  Interventions: Other: RIA harvesting group

INTERVENTIONS:
Other: RIA harvesting group — Subjects allocated to the RIA group will have the graft harvested in a standardized fashion using the technique described by Quintero et al. Briefly, the RIA device is a single-pass reamer that is connected to an aspirator and irrigator, allowing simultaneous reaming, irrigation, and aspiration of the contents of the femoral canal. RIA head size and tube length will be chosen based on preoperative templating of anteroposterior and lateral radiographs of the donor femur (a head size of 2mm larger than the inner cortical diameter at the isthmus of the femur will be selected). Fluoroscopic imaging will be used to confirm guidewire positioning and avoid eccentric reaming. Bone graft will be harvested from the central femoral canal and from each femoral condyle in 3 separate passes.
  Arms: RIA harvesting group
Other: AICBG harvesting group — Iliac crest bone graft will be harvested from the anterior iliac crest through an incision beginning 2cm posterior to the anterior superior iliac spine and carried posteriorly. A window will be made in the iliac crest and a curette will subsequently be used to harvest the cancellous bone. The incision will be closed in 3 layers. The infiltration of local anaesthetic will be at the discretion of the surgeon.
  Arms: AICBG harvesting group

SUMMARY:
The specific question the investigators will seek to answer is: can the Reamer Irrigator Aspirator (RIA) provide a bone graft source for the treatment of nonunions that is equally effective to Autogenous Iliac Crest Bone Graft (AICBG) while resulting in a decreased amount of post-operative pain and a lower rate of complications?

DETAILED DESCRIPTION:
All subjects will be pre-screened by the treating physician. Subjects who present with a nonunion of a long bone will be invited to speak to the research coordinator regarding the study. An internet based randomization system will be used to allocate subjects to treatment groups. Participating sites will be given a unique ID and password to log into the secure website and register their subject.

Treating physicians will use 1 of 2 bone graft harvesting methods in patients with a nonunion of a long bone requiring grafting. The first method involves harvesting bone graft from the iliac crest area. The second method involves using the RIA to harvest bone graft from the femoral canal. Clinical assessments will occur at the time of hospital admission (baseline), at post-op day 1, and then at 2 weeks, 6 weeks, 3 months, 6 month, 12 months and 24 months post-surgery.

Surgical procedure at the nonunion site will not be standardized as this will vary greatly. Surgeons may use bone graft substitutes at the recipient site at their discretion. We will however, standardize surgical techniques for harvesting of the graft from the donor site.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male or female, aged 18-65
* Subjects with a nonunion of a long bone requiring bone grafting in the -opinion of their orthopaedic surgeon (nonunion will be defined as "9 months duration of the nonunited fracture with no evidence of progressive healing over the previous 3 months")
* Subjects must have an uninjured, healthy iliac crest and a femur that has not previously been operated on
* Subjects must provide informed consent

Exclusion Criteria:

* Subjects requiring a structural bone graft
* Subjects presenting with an active systemic or local infection
* Subjects with a nonunion due to pathologic fracture
* Patients with severely compromised soft-tissue coverage at the nonunion site, sufficient to impair bone healing
* Patients receiving radiation, chemotherapy, immunosuppression, or chronic steroids
* Subjects with whom there are likely to be problems, in the judgment of the Investigator or Research Coordinator, with maintaining follow-up (such as no fixed address, plans to move out of town in the next year, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2012-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by a Visual Analog Scale (VAS) | 6 weeks post operatively
  Our primary outcome will be acute post-operative pain at the donor site, measured by a pain visual analog scale (VAS)at 6 weeks post-operatively

SECONDARY OUTCOMES:
Time to union | 1 year
  Secondary outcomes will include time to union,

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Nauth, MD FRCS(C), Principal Investigator — Unity Health Toronto
Locations (1):
- St.Michael's Hospital, Toronto, Ontario, Canada